CLINICAL TRIAL: NCT00248638
Title: Phase III Study on the Efficacy of Glutamine Dipeptide-Supplemented Parenteral Nutrition in Surgical ICU Patients
Brief Title: Efficacy and Mechanisms of GLN Dipeptide in the SICU
Acronym: GLND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thomas R. Ziegler, MD, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00024944; U01DK069322 (NIH); DK69322 (Other: Other); NCT01776476 (obsolete NCT alias)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glutamine dipeptide (Active Comparator): Glutamine dipeptide supplemented nutrition to be given to participants.
  Interventions: Drug: Glutamine dipeptide with 15% Clinisol
- standard (Placebo Comparator): Participants given standard nutrition without glutamine dipeptide
  Interventions: Drug: 15% Clinisol

INTERVENTIONS:
Drug: Glutamine dipeptide with 15% Clinisol — Subjects randomized to AG-PN will receive PN containing 0.5 g/kg/day of L alanyl L GLN (AG) dipeptide (Dipeptiven 20%; Fresenius-Kabi) and 1.0 g/kg/day of 15% Clinisol (Baxter Inc., Deerfield, IL) AA solution (total = 1.5 g/kg/day, with AG replacing 1/3 of Clinisol AA). The amount of GLN dipeptide administered each day will be determined by daily PN volume intake data.
  Other Names: Alanyl-glutamine Dipeptide; Dipeptiven
  Arms: Glutamine dipeptide
Drug: 15% Clinisol — Subjects randomized to STD-PN will receive 1.5 g/kg/day of 15% Clinisol. The amount of Clinisol administered each day will be determined by daily PN volume intake data.
  Arms: standard

SUMMARY:
Relative glutamine (GLN) deficiency may contribute to morbidity and mortality in surgical intensive care unit (SICU) patients. During critical illness, GLN utilization by the immune system, gut mucosa and other tissues exceeds endogenous production and plasma GLN concentrations decrease, which may contribute to cellular dysfunction and increase nosocomial infection risk and mortality. Conventional GLN-free parenteral nutrition (PN) has a limited impact on SICU outcomes and does not repair the GLN deficit. Recent pilot data show that GLN dipeptide-supplemented PN decreases nosocomial infections and improves clinical outcomes in SICU patients. The process of benefit is poorly understood, but animal and human data suggest that GLN treatment correlates with a) up-regulation of cytoprotective molecules in blood and tissues [e.g, GSH, specific heat shock proteins (HSPs) and GLN]; and b) improved epithelial barrier defenses and immune cell number and function. Properties of L-GLN limit provision in solution, but the GLN dipeptide alanyl-GLN (AG) confers stability and solubility in PN (AG-PN). Investigators propose a multicenter, double-blind, randomized, controlled phase III trial based on our pilot data to test the hypothesis that AG-PN improves clinical outcomes in SICU patients requiring PN after cardiac, vascular or colonic operations. Subjects will receive either standard GLN-free PN or isocaloric, isonitrogenous, AG-PN until enteral feeds are established. Specific Aim 1 is to determine whether AG-PN decreases hospital mortality, nosocomial infection and other important indices of morbidity. Specific Aim 2 is to obtain novel, mechanistically relevant observational data in the Aim 1 subjects on whether AG-PN a) increases serial blood levels of GSH, HSP-70 and -27, and GLN; b) decreases the presence in serum of the bacterial products flagellin and LPS and the adaptive immune response to these mediators; and c) improves key indices of innate/adaptive immunity. This study is designed to delineate the clinical benefit of a major new nutrition support strategy in high-risk SICU patients.

.

DETAILED DESCRIPTION:
Overview: Relative deficiency of glutamine (GLN) appears to contribute to morbidity and mortality in surgical intensive care unit (SICU) patients, but conventional nutrition support does not repair this deficit. GLN requirements increase during critical illness when utilization by the immune system, gut mucosa and other tissues exceeds endogenous production. GLN depletion under these conditions may contribute to hospital morbidity and mortality. Conventional parenteral nutrition (PN) does not contain GLN and thus does not prevent GLN depletion in catabolic patients. However, a pilot study and other reports strongly suggest that GLN-supplemented PN improves metabolic and clinical outcomes in critically ill patients. Underlying mechanisms for GLN action are poorly understood, but may involve systemic upregulation of the cytoprotective molecules glutathione (GSH), specific heat shock proteins (HSP) and GLN itself, improved gut barrier defenses, and improved innate and/or adaptive immune function. Properties of L-GLN limit provision in PN, but the dipeptide alanyl-glutamine (AG) confers stability and solubility in PN solutions. The pilot study demonstrated a marked decrease in nosocomial infection, improved indices of organ function, and a possible decrease in hospital mortality in SICU patients receiving AG-supplemented PN (AG-PN) versus standard, GLN-free PN (STD-PN). Investigators propose a multi-center, double-blind, controlled, Phase III trial, based on a pilot study, that will determine the effect of parenteral GLN on important clinical outcomes in patients requiring SICU care and PN after cardiac, vascular or colonic surgery. Investigators also propose to obtain needed hypothesis-generating, descriptive data from the Aim 1 study subjects to inform subsequent, truly mechanistic studies of GLN action in animal and human models of surgical critical illness. Study subjects will be randomized on an intent-to-treat basis to receive AG-PN or isonitrogenous, isocaloric STD-PN until enteral feeding is established.

Hypotheses:

1. SICU patients receiving PN supplemented with GLN dipeptide (AG-PN) will demonstrate improved clinical outcomes compared to patients receiving STD-PN.
2. Administration of AG-PN in the Aim 1 study subjects: a) increases serial blood levels of specific cytoprotective molecules and improves systemic redox status; b) is associated with decreased serum positivity for the bacterial products flagellin and lipopolysaccharide ( LPS) and the adaptive immune response to these mediators; and c) improves key indices of innate/adaptive immunity.

Specific Aims:

Aim 1: To perform a Phase III randomized controlled trial (RCT) to determine whether AG-PN decreases hospital mortality, nosocomial infections, and other indices of hospital morbidity versus STD-PN in SICU patients. The study will test whether AG-PN: decreases hospital mortality and the incidence of nosocomial infection (primary endpoints) in SICU patients after cardiac, vascular or colonic surgery. We will also determine whether AG-PN decreases total hospital infections, bloodstream infections (BSI), infections due to Staphylococcus aureus or fungal species, the number of days patients require mechanical ventilation, the SICU and total hospital length of stay and the 6-month mortality rate (secondary endpoints).

Aim 2: To determine in the Aim 1 study subjects whether AG-PN: a) increases systemic blood concentrations of the cytoprotective molecules GSH, HSP-70, HSP-27 and GLN and improves systemic GSH and cysteine redox status; b) is associated with decreased serum positivity for the bacterial products flagellin and LPS and titers of anti-flagellin and anti-LPS immunoglobulin M (IgM), immunoglobulin A (IgA) and immunoglobulin G (IgG); and c) improves key indices of innate/adaptive immune cell function.

ELIGIBILITY:
Inclusion criteria: 1) A signed informed consent is in place on the patient's chart; 2) The patient is at least 18 but not more than 90 years of age at time of surgery; 3) The patient has a body mass index (BMI) < 40 kg/m2 prior to surgery; 4) The patient currently requires SICU care and is within 14 days postoperative from one of the following open (non-laparoscopic) surgical procedures: coronary artery bypass graft(CABG), cardiac valve, vascular (non-neurosurgical), or esophageal gastrointestinal resection of esophagus, stomach, small bowel, colon and/or rectum), or operation to identify the source of peritonitis when there is evidence of a bowel perforation (with or without bowel resection); 5) The patient will require central venous PN for 7+ subsequent days after entry on a clinical basis≠; 6) There is central venous access for administration of the study PN; and 7) The patient's primary physician(s) will allow the investigative team to manage the study PN and enteral feedings during the current hospitalization.

Exclusion Criteria: 1) The patient is pregnant; 2) The patient has clinical sepsis [defined as unstable blood pressure despite pressor support AND mean arterial pressure (MAP) < 60 mm Hg on at least 3 consecutive readings within a 3-hour period during the 24 hours prior to study entry; 3) a) The patient has a current malignancy requiring surgery as the GLND qualifying operation OR b) the patient is currently receiving an active regimen of chemotherapy and/or radiotherapy to treat a previously diagnosed malignancy†; 4) The patient has a history of seizures or pre-existing seizure disorder; 5) The patient has a current encephalopathy*; 6) The patient has a known history of cirrhosis OR a serum total bilirubin level ≥ 10.0 mg/dL); 7) The patient has a history of chronic renal failure requiring dialysis, or has significant renal dysfunction (defined as serum creatinine > 2.5 mg/dL and is not receiving continuous renal replacement therapy (CRRT) or the patient requires acute hemodialysis postoperatively; 8) The patient has a concomitant burn or trauma injury; 9) The patient has previously undergone an organ transplantation;10) the patient has a history of HIV/AIDS; 11) The patient has received any investigational drug within 60 days prior to study entry; 12) The patient has received enteral or parenteral enteral feedings enriched in arginine and/or glutamine within 30 days prior to study entry; and 13) The patient is unable or unwilling to participate in study procedures such as longitudinal blood draws and out patient follow-up visits, etc.

*Encephalopathy for GLND can be diagnosed only in non-chemically sedated patients by the primary critical care physicians or neurologist consultants and is defined as either a comatose state OR severe abnormalities diagnosed by electroencephalogram (EEG), OR if all of the following criteria are met: a) patient goes to sleep but is arousable to verbal and painful stimuli; does not open eyes spontaneously (decreased level of consciousness); b) patient exhibits severe confusion or complete disorientation when aroused (disorientation); c) patient exhibits severe lethargy or bizarre behavior (behavioral dysfunction); and d) patient exhibits inability to cooperate, asterixis, ataxia, clonus, decortication, decerebration, seizures, or rigidity (severe neuromuscular dysfunction).

† Patients with malignant metastasis and terminal untreatable carcinoma will be excluded as per the operational definition agreed upon by the Data Safety and Monitoring Board (DSMB).

≠ Please note that the patient should be in the SICU at the initial PN hang time.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Ziegler, MD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - The Miriam Hospital/Brown University, Providence, Rhode Island
  - Vanderbilt University, Nashville, Tennessee
  - University Of Wisconsin Hospital, Madison, Wisconsin

REFERENCES:
- [Derived] Ziegler TR, May AK, Hebbar G, Easley KA, Griffith DP, Dave N, Collier BR, Cotsonis GA, Hao L, Leong T, Manatunga AK, Rosenberg ES, Jones DP, Martin GS, Jensen GL, Sax HC, Kudsk KA, Galloway JR, Blumberg HM, Evans ME, Wischmeyer PE. Efficacy and Safety of Glutamine-supplemented Parenteral Nutrition in Surgical ICU Patients: An American Multicenter Randomized Controlled Trial. Ann Surg. 2016 Apr;263(4):646-55. doi: 10.1097/SLA.0000000000001487. PMID 26501700

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glutamine Dipeptide | Standard
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adults following CABG, cardiac valve, vascular (non-neurosurgical), or small bowel and/or colonic surgery who are deemed likely to require PN for ≥ 7 subsequent days by the attending physicians and investigators are eligible. Potentially eligible subjects admitted to the SICU and deemed to require PN.
Groups:
- Total: Total of all reporting groups
Arm/Group | Glutamine Dipeptide | Standard | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 50 | 93
  >=65 years | 32 | 25 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (13.6) | 60.4 (13.0) | 60.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 30 | 70
  Male | 35 | 45 | 80
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Hospital Mortality Rate
Description: Number of participants who died during hospitalization.
Time Frame: Current Hospitalization (Up to 6 Months)
Measure: Number; unit: participants
Arm/Group | Glutamine Dipeptide | Standard
Number analyzed (Participants) | 75 | 75
participants | 11 | 13

2. Primary Outcome: Percentage of Patients Who do Not Develop Hospital Infections
Description: Subjects remaining infection-free during the hospitalization.
Time Frame: Current Hospitalization (Up to 6 Months)
Measure: Number; unit: percentage of participants
Groups:
- Glutamine Dipeptide: Glutamine dipeptide supplemented nutrition to be given to participants.
  Glutamine dipeptide: Subjects randomized to AG-PN will receive PN containing 0.5 g/kg/day of L alanyl L GLN (AG) dipeptide (Dipeptiven 20%; Fresenius-Kabi) and 1.0 g/kg/day of 15% Clinisol (Baxter Inc., Deerfield, IL) AA solution (total = 1.5 g/kg/day, with AG replacing 1/3 of Clinisol AA). Subjects randomized to STD-PN will receive PN AA as the standard, GLN-free amino acid solution (15% Clinisol). The AA solutions are nearly isonitrogenous; STD-PN provides 2.35 g nitrogen and the AG-PN provides 2.45 g nitrogen per 100 ml 15% AA solution. The amount of GLN dipeptide administered each day will be determined by daily PN volume intake data.
  Study subjects will receive a maximum of 28 days of study PN (blinded placebo or GLN-dipeptide-supplemented PN). If the subject continues to require PN after Day 28, study PN and GLN dipeptide will be discontinued.
- Standard: Participants given standard nutrition without glutamine dipeptide
  Glutamine dipeptide: Subjects randomized to AG-PN will receive PN containing 0.5 g/kg/day of L alanyl L GLN (AG) dipeptide (Dipeptiven 20%; Fresenius-Kabi) and 1.0 g/kg/day of 15% Clinisol (Baxter Inc., Deerfield, IL) AA solution (total = 1.5 g/kg/day, with AG replacing 1/3 of Clinisol AA). Subjects randomized to STD-PN will receive PN AA as the standard, GLN-free amino acid solution (15% Clinisol). The AA solutions are nearly isonitrogenous; STD-PN provides 2.35 g nitrogen and the AG-PN provides 2.45 g nitrogen per 100 ml 15% AA solution. The amount of GLN dipeptide administered each day will be determined by daily PN volume intake data.
  Study subjects will receive a maximum of 28 days of study PN (blinded placebo or GLN-dipeptide-supplemented PN). If the subject continues to require PN after Day 28, study PN and GLN dipeptide will be discontinued.
Arm/Group | Glutamine Dipeptide | Standard
Number analyzed (Participants) | 75 | 75
percentage of participants | 56 | 69

3. Secondary Outcome: Mean Glutathione Level
Description: Glutathione (GSH) levels will be measured in µM (micro moles) from baseline to day 28. Higher levels indicate a higher GSH presence.
Time Frame: Baseline, Day 3, Day 7, Day 14, Day 21, Day 28
Population: The number of participants currently hospitalized are included in each time point analysis.
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Glutamine Dipeptide | Standard
Number analyzed (Participants) | 75 | 75
µM
  Baseline: number analyzed (Participants) | 53 | 54
  Baseline | 1.850 (.195) | 1.880 (.182)
  Day 3: number analyzed (Participants) | 46 | 47
  Day 3 | 1.524 (.156) | 1.374 (.162)
  Day 7: number analyzed (Participants) | 42 | 43
  Day 7 | 5.056 (3.619) | 1.473 (.202)
  Day 14: number analyzed (Participants) | 32 | 31
  Day 14 | 1.312 (.220) | 1.327 (.306)
  Day 21: number analyzed (Participants) | 20 | 24
  Day 21 | 1.286 (.266) | 1.597 (.297)
  Day 28: number analyzed (Participants) | 20 | 21
  Day 28 | 1.279 (.232) | 1.430 (.301)

4. Secondary Outcome: Mean Heat Shock Proteins Level, HSP70
Description: Levels of the heat shock protein,HSP70, will be measured in ng/mL from baseline to day 28. Higher levels indicate a higher protein presence.
Time Frame: Baseline, Day 3, Day 7, Day 14, Day 21, Day 28
Population: The number of participants currently hospitalized are included in each time point analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Glutamine Dipeptide | Standard
Number analyzed (Participants) | 75 | 75
ng/mL
  Baseline: number analyzed (Participants) | 74 | 72
  Baseline | 52.6 (6.2) | 55.3 (8.7)
  Day 3: number analyzed (Participants) | 72 | 67
  Day 3 | 48.1 (6.0) | 44.5 (5.8)
  Day 7: number analyzed (Participants) | 67 | 64
  Day 7 | 52.1 (7.0) | 36.4 (3.1)
  Day 14: number analyzed (Participants) | 48 | 39
  Day 14 | 33.9 (4.6) | 33.9 (4.0)
  Day 21: number analyzed (Participants) | 33 | 31
  Day 21 | 30.7 (4.0) | 32.9 (6.7)
  Day 28: number analyzed (Participants) | 29 | 24
  Day 28 | 26.3 (3.1) | 25.5 (3.7)

5. Secondary Outcome: Mean Heat Shock Proteins Level, HSP27
Description: Levels of the heat shock protein, HSP27, will be measured in pg/mL from baseline to day 28. Higher levels indicate a higher protein presence.
Time Frame: Baseline, Day 3, Day 7, Day 14, Day 21, Day 28
Population: The number of participants currently hospitalized are included in each time point analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Glutamine Dipeptide | Standard
Number analyzed (Participants) | 75 | 75
pg/mL
  Baseline: number analyzed (Participants) | 74 | 72
  Baseline | 1171.1 (70.9) | 1134.3 (76.0)
  Day 3: number analyzed (Participants) | 72 | 67
  Day 3 | 1189.3 (68.9) | 1140.0 (71.1)
  Day 7: number analyzed (Participants) | 67 | 64
  Day 7 | 1222.4 (82.0) | 1259.0 (91.5)
  Day 14: number analyzed (Participants) | 48 | 39
  Day 14 | 1161.0 (98.7) | 1253.4 (107.1)
  Day 21: number analyzed (Participants) | 33 | 31
  Day 21 | 1314.3 (119.7) | 1250.9 (163.2)
  Day 28: number analyzed (Participants) | 29 | 23
  Day 28 | 1177.5 (137.8) | 880.9 (144.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout each participant's hospital stay (up to six months).
Arm/Group | Glutamine Dipeptide | Standard
All-Cause Mortality (participants affected / at risk) | 11/75 | 13/75
Serious Adverse Events (participants affected / at risk) | 39/75 | 40/75
Other Adverse Events (participants affected / at risk) | 22/75 | 12/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glutamine Dipeptide (N=75) | Standard (N=75)
death (General disorders) | 15 (15) | 19 (19)
rehospitalization (Surgical and medical procedures) | 15 (16) | 13 (15)
re-operation within 30 days (Surgical and medical procedures) | 16 (30) | 14 (28)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glutamine Dipeptide (N=75) | Standard (N=75)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 11 (14)
tracheostomy (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 12 (12)
significant bleeding (General disorders) | 9 (11) | 6 (7)
ICU readmission (General disorders) | 14 (16) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No